CLINICAL TRIAL: NCT06407817
Title: Comparative Effects Of Spencer and Reverse Distraction Technique In Patients With Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0184
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spencer's technique (Experimental): This group will receive the Spencer's technique.
  Interventions: Procedure: Spencer technique; Procedure: reverse distraction technique
- reverse distraction technique (Active Comparator): This group will recieve reverse distraction technique
  Interventions: Procedure: Spencer technique; Procedure: reverse distraction technique

INTERVENTIONS:
Procedure: Spencer technique — No of repetitions; 3 sets for 10 repetitions with 1 minute rest between sets No Of Sessions Per Week: 3 Per Weeks for 6 weeks (40 Min per Session)
Procedure: reverse distraction technique — No of repetitions; 10 ( Shoulder Abduction)10 ( Shoulder Flexion) 10 (Shoulder External Rotation) No Of Sessions Per Week: 3 Per Weeks for 6 weeks (40 Min Per Session)

SUMMARY:
To compare the effects of spencer and reverse distraction technique in patients with adhesive capsulitis

DETAILED DESCRIPTION:
Adhesive capsulitis, also known as frozen shoulder, is an inflammatory condition characterized by shoulder stiffness, pain, and significant loss of passive range of motion. Adhesive capsulitis has a prevalence of approximately 2% to 5% in the general population, with a mean onset of age of 55.

A randomized clinical trial will be conducted at Ibne Sina Hospital, Multan . Non probability convenience sampling technique will be applied on 50 patients who will be allocated through computerized randomization into group A & group B to collect data. Group A will be given spencer technique and group B will be given reverse distraction technique along with baselines. The study will be completed within the time duration of ten months. Primary Outcome measures of the research will be pain, range of motion, function, muscle strength, disability and quality of life will be measured pre and post intervention. The whole treatment protocols will be given for four weeks. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age group 40-60 years
* Male and female
* Positive Capsular pattern (ER more limited than Abd which is more limited than IR)
* Limitation in shoulder ROM ; Flexion <180 , Abduction <180 , External Rotation <50
* Patients of stage 2 and 3 of adhesive capsulitis

Exclusion Criteria:

* History of surgery of the affected shoulder
* Fractures in around the shoulder
* Neurological disorders leading to altered muscle activity
* Systemic arthritic conditions (RA, Osteoporosis)
* Disorders of the cervical spine

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
pain : numerical pain rating scale | 6 weeks
  Patients' overall assessment of pain will be provided using the numeric pain rating scale (NPRS). The NPRS is known to be a sensitive and reliable scale for clinical and experimental evaluation of pain intensity. The score ranges from 0, indicating no pain, to 10, expressing worst imaginable pain. The reliability of numeric pain rating scale (NPRS) is 0.92 (0.87, 0.95).
range of motion : universal goniometer | 6 weeks
  Universal Goniometer is the most commonly utilised clinical tool for measuring joint range of motion due to its ease of use, low cost, and demonstrated reasonable levels of reliability and validity in numerous studies. Validity and intertester reliability (r =.97-.98; ICC =.98-.99) are both high
shoulder pain and impairment : SPADI | 6 weeks
  The SPADI consists of 13 items that assess two domains: a 5-item subscale for pain and an 8-item subscale for disability. The SPADI has since been used in both primary care on mixed diagnosis and surgical patient populations including rotator cuff disease, osteoarthritis, and rheumatoid arthritis, adhesive capsulitis ,joint replacement surgery , and in a large population-based study of shoulder symptoms (37).
  Reliability- 0.89, Validity - 0.90
36-Item Short Form Health Survey questionnaire (SF-36) | 6 weeks
  The 36-Item Short Form Health Survey questionnaire (SF-36) is a very popular instrument for evaluating Health-Related Quality of Life. The ICC for SF-36 PF is (0.96, 95% CI 0.92-0.98) so it's a reliable test.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University
Locations (1):
- Johar Pain Relief Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No